CLINICAL TRIAL: NCT06381401
Title: The Efficacy of Bupivacaine 0.125% Versus Bupivacaine 0.25% in Superficial Cervical Plexus Block on Operative Field Visibility for Adults Undergoing Tympanomastoid Surgeries, A Prospective Randomized Controlled Study
Brief Title: Bupivacaine 0.125% Versus Bupivacaine 0.25% in Superficial Cervical Plexus Block for Tympanomastoid Surgeries in Adults
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS-492-2023
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Surgical Field; Acute Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine 0.25% (Active Comparator): Patients will receive superficial cervical plexus block using 0.25% bupivacaine (5ml of bupivacaine 0.5% + 5ml normal saline).
  Interventions: Drug: bupivacaine 0.25%
- Bupivacaine 0.125% (Active Comparator): Patients will receive superficial cervical plexus block using 0.125% bupivacaine (2.5ml of bupivacaine 0.5% + 7.5ml normal saline).
  Interventions: Drug: bupivacaine 0.125%

INTERVENTIONS:
Drug: bupivacaine 0.25% — superficial cervical plexus block using 10 ml of bupivacaine 0.25%
  Arms: Bupivacaine 0.25%
Drug: bupivacaine 0.125% — superficial cervical plexus block using 10 ml of bupivacaine 0.125%
  Arms: Bupivacaine 0.125%

SUMMARY:
Bleeding is one of the most common complications in tympanomastoid surgery that could prolong the time of operation and also might lead to morbidity. Pain is also one of the most annoying complications of tympanomastoid surgeries. Thus, adequate surgical field visualization is utmost important. A bloodless field allows optimal exposure and identification of vital neurovascular structures. Even small bleeding, inconsequential for the patient's volume status, can create great technical difficulty in the confined space of the tympan, leading to prolonged surgery, incomplete procedures, and increased complications.

The use of regional nerve blocks as an alternative to hypotensive anesthesia has gained popularity in recent years. The superficial cervical plexus block (SCPB) provides effective analgesia and reduces sympathetic activity, resulting in reduced bleeding and improved surgical conditions. The superficial cervical plexus (SCP) provides sensory innervation to the ear and surrounding structures, reducing pain perception during and after surgery.

This is the first randomized controlled clinical trial investigating the effect of combined general anesthesia with SCPB using 0.125% versus 0.25% bupivacaine during tympanomastoid surgery.

This study aims to compare the efficacy of two different concentrations of bupivacaine 0.125% & 0.25% in Superficial Cervical Plexus Block in patients undergoing tympanomastoid surgery on operative field visualization, intraoperative hemodynamic stability, and postoperative analgesia.

The investigators hypothesize that bupivacaine 0.125% would be non-inferior to bupivacaine 0.25% in achieving optimal surgical field visualization, hemodynamic stability, surgeon satisfaction and postoperative analgesia.

This prospective double-blinded study will be carried out on 60 patients between 21 to 70 years, with ASA I-II and undergoing tympanomastoid surgery. Participants were equally divided into two groups: Group A: Patients received SCPB using 0.25% bupivacaine (5ml of bupivacaine 0.5% + 5ml normal saline). Group B: Patients received SCPB using 0.125% bupivacaine (2.5ml of bupivacaine 0.5% + 7.5ml normal saline).

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 21 - 70 years.
2. Patients undergoing tympanomastoid surgery.
3. Both genders.
4. ASA physical class I and II.

Exclusion Criteria:

1. Patient refusal.
2. Uncooperative patients.
3. Allergy to the drug enrolled in the study.
4. Anatomical abnormality at injection site.
5. Infection at injection site.
6. Bleeding disorders.
7. ASA physical class III and IV patients.
8. Patients having significant chronic diseases as: uncontrolled asthma, cardiovascular disorders (significant arrhythmias, severe valvular diseases, congenital heart diseases, ischemic heart disease, or cardiomyopathy).
9. Renal impairment (creatinine level ≥ 2mg/dl), or uncompensated chronic liver disease.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
The total consumption of IV glyceryl trinitrate | up to 5 hours
  The total consumption of IV glyceryl trinitrate administered to maintain a surgical field with a Boezaart bleeding score ≤2 (grade 0 = no bleeding, grade 5 = severe bleeding threatening surgical field)

SECONDARY OUTCOMES:
Fentanyl consumption | up to 5 hours
  Total intraoperative consumption of fentanyl
Postoperative pain | 1 hour postoperatively
  Postoperative pain is measured by Visual Analog Scale (0 = no pain, 10 = worst imaginable pain)
Postoperative hospital stay | 4 days
  Duration of postoperative hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Nevan M Mekawy, M.D., Study Chair — Professor of Anesthesiology, Surgical ICU & Pain Management, Cairo University; Mohsen M Waheb, M.D., Study Director — Lecturer of Anesthesiology, Surgical ICU & Pain Management, Cairo University; Kareem MA Nawwar, M.D., Study Director — Lecturer of Anesthesiology, Surgical ICU & Pain Management, Cairo University; Fatma A Mohamed Hassan, M.B.B.Ch., Principal Investigator — Resident of Anesthesia, Surgical ICU & Pain Management
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt